CLINICAL TRIAL: NCT06475937
Title: A Phase I, Multicenter, Open-label, First-in-Human, Dose Escalation and Expansion Study of DM001 in Patients With Advanced Solid Tumors
Brief Title: A Study of DM001 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xadcera Biopharmaceutical (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Doma Biopharmaceutical（Suzhou）Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM001001
Record Dates: First submitted 2024-06-07; First posted 2024-06-26 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-02

CONDITIONS: Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Solid Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DM001 administrated to subjects with advanced or metastatic solid tumors (Experimental): An IV infusion of DM001 will be administrated approximately 30-60 min on Day 1 once Q3W
  Interventions: Drug: DM001

INTERVENTIONS:
Drug: DM001 — Subjects may continue to receive DM001 (with an increased dose that has been assessed as safe in the dose-escalation period) once every 3 weeks (Q3W) for a total of 6 cycles at the discretion of the investigators, until unacceptable toxicity, progressive disease (PD), or withdrawal of consent.

SUMMARY:
The goal of this clinical trial is to find out about the safety, efficacy, and tolerability of DM001 for patients with the advanced solid tumors. DM001 is an experimental drug which is not approved by health authorities for the treatment of advanced solid tumors.

Participants will have up to 17 visits during the study.There will be up to a 4-week Screening Period followed by a treatment period that will be divided into 3-week cycles/ Participants will have 5 study visits during Cycle 1, 3 visits during Cycles 2 and 3, and 1 visit during subsequent cycles. Participants will have an End of Treatment visit 21 days (+ 7 days) after last dose of study drug and then a follow-up visit 30 days (± 7 days) after the End of Treatment visit.

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, openlabel, first-in-human (FIH), doseescalation and dose expansion study to evaluate the safety, tolerability, PK, and preliminary efficacy of DM001 in subjects with advanced solid tumors.

DM001, a bispecific ADC developed using fully human antibodies with a common light chain, which targets TROP2 and EGFR.

DM001 is sterile yellowish-green lyophilized powder for IV infusion.

Subjects with solid malignant tumors will be treated with DM001 on Day 1 once Q3W (dose adjustments may be required depending on the safety profile and PK data of each dose).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have the ability to understand and willingness to sign a written informed consent document.
2. Subjects who have pathologically or cytologically confirmed documented metastatic/advanced breast cancer, EGFRmut or EGFRwt NSCLC, gastric cancer, gastroesophageal cancer or CRC, and have progressed on standard therapy, or intolerant to standard therapy, or no standard therapy accessible to the subjects due to any reason.
3. Subjects must be ≥18 years of age at the time of signing the informed consent form.
4. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Has a life expectancy of ≥3 months.
6. Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

Exclusion Criteria:

1. Subjects have another active invasive malignancy within 5 years.
2. Current or history of a hematologic malignancy.
3. Primary central nervous system (CNS) malignancies or CNS metastases. Individuals with brain metastases can be enrolled only if treated, nonprogressive brain metastases and off high-dose steroids (>20 mg prednisone or equivalent) for at least 4 weeks.
4. Individuals with Gilbert's disease with ≥3 × ULN.
5. Has an uncontrolled infection requiring intravenous (IV) injection of antibiotics, antivirals, or antifungals.
6. Has a medical history of clinically significant lung diseases or is suspected to have these diseases by imaging at the screening period.
7. Clinically uncontrolled intercurrent illness, including but not limit to an ongoing active infection, active coagulopathy, uncontrolled cardiovascular disease, uncontrolled immune disease, uncontrolled diabetes, uncontrolled pleural and peritoneal effusion, psychiatric illness that would limit compliance with the study requirements and other serious medical illnesses requiring systemic therapies.
8. Mean resting corrected QT interval corrected by Fridericia's formula (QTcF, QTcF=QT/[RR]1/3) >470 msec obtained from triplicate 12-lead ECGs at baseline; no concomitant medications that would prolong the QT internal; no family history of long QT syndrome.
9. Known human immunodeficiency virus infection, or active hepatitis B virus (HBV), or hepatitis C virus (HCV) infection. Chronic carriers of HBV infection (hepatitis B surface antigen-positive, undetectable, or low HBV DNA) who receive prophylactic treatment during the study can be enrolled. Subjects with a history of HCV infection have completed curative antiviral treatment and HCV viral load below the limit of quantification and HCV antibody positive but HCV RNA negative due to prior treatment or natural resolution should be eligible.
10. Females who are pregnant or lactating or who intend to become pregnant during participation in the study are not eligible to participate.
11. Subjects who are of reproductive potential refuse to use effective methods of birth control during the course of participation in the study and within 120 days for both women and men of the last dose are ineligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-08-13 (Estimated); Study Completion 2027-02-13 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicities (DLTs) of DM001 | 12 months
  Incidence of DLTs of DM001 will be determined. A dose-limiting toxicity (DLT) was defined as grade 3 neurological toxicities (e.g. chemical meningitis) or other grade 4 toxicity.
Maximum tolerated dose (MTD) for DM001 | 12 months
  The MTD of DM001 will be determined. The MTD was defined as the dose where 0/3 or 1/6 patients experienced a DLT with at least two patients encountering DLT at the higher dose.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC(0-inf), ng*h/mL) | 12 months
  Area under the plasma concentration-time curve from time zero extrapolated to infinity, calculated by linear up/log down trapezoidal summation.
Maximum (peak) plasma concentration (Cmax, ng/mL) | 12 months
  Maximum concentration, obtained directly from the observed concentration versus time data.
Time to maximum (peak) concentration (Tmax, h) | 12 months
  Time to Cmax
Trough concentration (Ctrough, ng/mL) | 12 months
  The lowest plasma concentration reached before the next dose.
Objective response rate (ORR) | 12 months
  ORR is defined as the number of patients with at least a confirmed complete response (CR) or partial response (PR), based on the best objective response values while on treatment using RECIST version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Zhaorong Chen, CMO, Study Chair — Xadcera Biopharmaceutical (Suzhou) Co., Ltd.
Locations (5):
- United States (2):
  - Sarah Cannon Research Institute (SCRI), Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Icon Cancer Centre South Brisbane, South Brisbane, Queensland
  - Tasman Oncology Research, Southport, Queensland
  - Monash Health, Clayton, Victoria